CLINICAL TRIAL: NCT02581410
Title: Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Adults ≥ 65 Years of Age With and Without Zostavax® Vaccination at Least 5 Years Earlier
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Herpes Zoster Subunit (HZ/su) Vaccine (GSK1437173A) in Adults ≥ 65 Years of Age With and Without Zostavax® Vaccination at Least 5 Years Earlier
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201198
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Results first posted 2017-09-26 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Herpes Zoster
Keywords: Zostavax®; ≥ 65 years of age; Herpes Zoster; Shingles; Immunogenicity; Safety
MeSH Terms: conditions — Herpes Zoster | interventions — Vaccines

ARMS (2):
- GSK1437173A Group (Experimental): Subjects ≥ 65 years of age who received Zostavax vaccine ≥ 5 years earlier and received 2 doses of the HZ/su vaccine (first dose given at Month 0 and second dose given 2 months later) in this study.
  Interventions: Biological: GSK Biologicals Herpes Zoster subunit (HZ/su) vaccine (GSK 1437173A)
- Control Group (Active Comparator): Subjects ≥ 65 years of age who never received Zostavax vaccine and received 2 doses of the HZ/su vaccine (first dose given at Month 0 and second dose given 2 months later) in this study.
  Interventions: Biological: GSK Biologicals Herpes Zoster subunit (HZ/su) vaccine (GSK 1437173A)

INTERVENTIONS:
Biological: GSK Biologicals Herpes Zoster subunit (HZ/su) vaccine (GSK 1437173A) — 2 doses administered by intramuscular (IM) injection into the deltoid muscle of the non-dominant arm.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of GSK Biologicals' HZ/su vaccine in adults ≥ 65 years of age with and without Zostavax® vaccination at least 5 years earlier.

DETAILED DESCRIPTION:
The study will evaluate two parallel groups of 200 adults ≥ 65 YOA; one group (Prev-Zvax) with a previous Zostavax® vaccination at least 5 years earlier, versus the other group without a previous Zostavax® vaccination (No prev-Zvax). The goal of this study is to generate immunogenicity, safety and reactogenicity data for the respective vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female ≥ 65 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject prior to performing any study specific procedure.

For the No prev-Zvax group only:

• No previous vaccination with Zostavax.

For the Prev-Zvax group only:

• Previous vaccination with Zostavax ≥ 5 calendar years earlier.

* Documentation indicating the date of previous Zostavax vaccination will be required.

Exclusion Criteria:

* Previous vaccination with Zostavax < 5 calendar years earlier and/or anyone that ever received more than a single dose of Zostavax.
* Previous vaccination against VZV, administration of HZ/su vaccine or any other investigational or non-registered HZ vaccine (except Zostavax for the Prev-Zvax group).
* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as > 14 consecutive days) of immunosuppressants or other immune-modifying drugs in the period starting 6 months prior to the first dose of vaccine. (For corticosteroids, a prednisone dose of < 20 mg/day, or equivalent, is allowed.) Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration of long-acting immune-modifying drugs (e.g., infliximab) in the period starting 6 months prior to the first vaccine dose or expected administration at any time during the study period.
* Administration or planned administration of a live vaccine in the period starting 30 days before the first dose of study vaccine and ending 30 days after the last dose of study vaccine, or, administration or planned administration of a non-replicating vaccine in the period starting 8 days prior to and ending 14 days after either dose of study vaccine.
* Current participation in or planned concurrent participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Planned administration of an HZ vaccine (including an investigational or non-registered vaccine) other than the study vaccine during the entire study.
* History of HZ or any suspected HZ between the screening visit and Visit 1.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine/product.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease (e.g., malignancy, human immunodeficiency virus [HIV] infection) or immunosuppressive/cytotoxic therapy (e.g., medications used during cancer chemotherapy, organ transplantation or to treat autoimmune disorders).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C (99.5°F) by oral route, axillary or tympanic setting, or ≥ 38.0°C/100.4°F on rectal setting. The recommended route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products in the period starting 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Significant underlying illness that, in the opinion of the investigator, would be expected to prevent completion of the study.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* Any condition which, in the judgment of the investigator, would make intramuscular (IM) injection unsafe.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 430 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (30):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Los Gatos, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Marlborough, Massachusetts
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Eau Claire, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Dagnew AF, Klein NP, Herve C, Kalema G, Di Paolo E, Peterson J, Salaun B, Schuind A. The Adjuvanted Recombinant Zoster Vaccine in Adults Aged >/=65 Years Previously Vaccinated With a Live-Attenuated Herpes Zoster Vaccine. J Infect Dis. 2021 Oct 13;224(7):1139-1146. doi: 10.1093/infdis/jiaa083. PMID 32103273
- [Derived] Grupping K, Campora L, Douha M, Heineman TC, Klein NP, Lal H, Peterson J, Vastiau I, Oostvogels L. Immunogenicity and Safety of the HZ/su Adjuvanted Herpes Zoster Subunit Vaccine in Adults Previously Vaccinated With a Live Attenuated Herpes Zoster Vaccine. J Infect Dis. 2017 Dec 12;216(11):1343-1351. doi: 10.1093/infdis/jix482. PMID 29029122
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 201198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 201198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 201198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK1437173A Group: Subjects above or equal to (≥) 65 years of age who received Zostavax vaccine ≥ 5 years earlier and received 2 doses of the GSK1437173A vaccine (first dose given at Month 0 and second dose given at Month 2) in this study.
- Control Group: Subjects ≥ 65 years of age who never received Zostavax vaccine and received 2 doses of the GSK1437173A vaccine (first dose given at Month 0 and second dose given at Month 2).in this study.
Period: Vaccination Phase
Arm/Group | GSK1437173A Group | Control Group
Started | 215 | 215
Completed | 213 | 212
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Migrated/moved from study area | 0 | 1
Period: End of Study Phase
Arm/Group | GSK1437173A Group | Control Group
Started | 215 | 215
Completed | 210 | 204
Not Completed | 5 | 11
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Migrated/moved from study area | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other-transfer of subject not completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GSK1437173A Group: Subjects ≥ 65 years of age who received Zostavax vaccine ≥ 5 years earlier and received 2 doses of the GSK1437173A vaccine (first dose given at Month 0 and second dose given at Month 2) in this study.
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Group | Control Group | Total
Number analyzed (Participants) | 215 | 215 | 430
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (4.5) | 70.8 (4.6) | 70.9 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 111 | 220
  Male | 106 | 104 | 210
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage: White - Caucasian / European Heritage | 215 | 215 | 430

OUTCOME MEASURES:

1. Primary Outcome: Anti-glycoprotein E (Anti-gE) Antibody (Ab) Concentrations
Description: Varicella Zoster Virus (VZV) gE Ab.Immunoglobulin G (IgG) was determined by Enzyme Linked Immunosorbent Assay (ELISA). Concentrations are presented as geometric mean concentrations (GMCs), expressed in milliinternational units per millilitre (mIU/mL). Geometric mean antibody concentrations were adjusted for group-matching variable.
Time Frame: One month after dose 2, at Month 3
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available at Month 3.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Groups:
- Control Group: Subjects ≥ 65 years of age who never received Zostavax vaccine and received 2 doses of the GSK1437173A vaccine (first dose given at Month 0 and second dose given at Month 2) in this study.
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 204 | 204
mIU/mL | 50522.9 [44347.4 to 57558.4] | 48589.4 [42649.4 to 55356.6]
Statistical Analysis 1: Comparison: GSK1437173A Group vs Control Group; To compare humoral immune responses at 1 month after dose 2 of GSK1437173A (Month 3) in subjects ≥ 65 years of age who received Zostavax ≥ 5 years earlier (Prev-Zvax) as compared to subjects who have never received Zostavax (No prev-Zvax); Test type: Non-Inferiority — Non-inferiority will be demonstrated if the upper limit of the two-sided 95% confidence interval of the adjusted geometric mean concentration (GMC) ratio (No prev- Zvax over Prev-Zvax) 1 month post-dose 2 is below 1.5 in terms of anti-gE antibodies; ANCOVA; Adjusted GMC ratio = 1.04, 95% CI 2-sided [0.92 to 1.17]

2. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = Occurrence of the symptom regardless of its intensity grade. Grade 3 pain = Significant pain at rest that prevented normal everyday activities. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) period after each dose.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 215 | 214
Participants
  Any Pain, Dose 1 | 171 | 159
  Grade 3 Pain, Dose 1 | 8 | 7
  Any Redness, Dose 1 | 69 | 48
  Grade 3 Redness, Dose 1 | 3 | 2
  Any Swelling, Dose 1 | 29 | 21
  Grade 3 Swelling, Dose 1 | 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 208 | 211
  Any Pain, Dose 2 | 163 | 161
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Pain, Dose 2 | 5 | 10
  Any Redness, Dose 2: number analyzed (Participants) | 208 | 211
  Any Redness, Dose 2 | 69 | 53
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Redness, Dose 2 | 6 | 2
  Any Swelling, Dose 2: number analyzed (Participants) | 208 | 211
  Any Swelling, Dose 2 | 29 | 27
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Swelling, Dose 2 | 0 | 1

3. Primary Outcome: Number of Days With Solicited Local Symptoms
Description: Solicited local symptoms were assessed during the 7-day (Days 0-6) period after each dose.
Time Frame: During the 7-day (Days 0-6) period after each dose.
Population: The analysis was performed on subjects with solicited local symptoms from the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and who had their symptom sheets filled in.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 171 | 161
Days
  Any Pain, Dose 1: number analyzed (Participants) | 171 | 159
  Any Pain, Dose 1 | 3.0 [2.0 to 4.0] | 2.0 [2.0 to 3.0]
  Any Redness, Dose 1: number analyzed (Participants) | 69 | 48
  Any Redness, Dose 1 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 4.0]
  Any Swelling, Dose 1: number analyzed (Participants) | 29 | 21
  Any Swelling, Dose 1 | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 4.0]
  Any Pain, Dose 2: number analyzed (Participants) | 163 | 161
  Any Pain, Dose 2 | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0]
  Any Redness, Dose 2: number analyzed (Participants) | 69 | 53
  Any Redness, Dose 2 | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 5.0]
  Any Swelling, Dose 2: number analyzed (Participants) | 29 | 27
  Any Swelling, Dose 2 | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0]

4. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (included nausea, vomiting, diarrhea and/or abdominal pain), headache, myalgia, shivering and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)] . Any = Occurrence of the symptom regardless of its intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) period after each dose.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 215 | 214
Participants
  Any Fatigue, Dose 1 | 69 | 59
  Grade 3 Fatigue, Dose 1 | 4 | 4
  Related Fatigue, Dose 1 | 62 | 48
  Any Gastro. int., Dose 1 | 31 | 14
  Grade 3 Gastro. int., Dose 1 | 2 | 2
  Related Gastro. int., Dose 1 | 24 | 9
  Any Headache, Dose 1 | 41 | 44
  Grade 3 Headache, Dose 1 | 4 | 1
  Related Headache, Dose 1 | 34 | 34
  Any Myalgia, Dose 1 | 47 | 42
  Grade 3 Myalgia, Dose 1 | 2 | 5
  Related Myalgia, Dose 1 | 41 | 37
  Any Shivering, Dose 1 | 25 | 17
  Grade 3 Shivering, Dose 1 | 2 | 1
  Related Shivering, Dose 1 | 22 | 16
  Any Fever, Dose 1 | 15 | 17
  Grade 3 Fever, Dose 1 | 0 | 0
  Related Fever, Dose 1 | 12 | 14
  Any Fatigue, Dose 2: number analyzed (Participants) | 208 | 211
  Any Fatigue, Dose 2 | 91 | 93
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Fatigue, Dose 2 | 9 | 11
  Related Fatigue, Dose 2: number analyzed (Participants) | 208 | 211
  Related Fatigue, Dose 2 | 85 | 84
  Any Gastro. int., Dose 2: number analyzed (Participants) | 208 | 211
  Any Gastro. int., Dose 2 | 30 | 27
  Grade 3 Gastro. int., Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Gastro. int., Dose 2 | 0 | 0
  Related Gastro. int., Dose 2: number analyzed (Participants) | 208 | 211
  Related Gastro. int., Dose 2 | 30 | 22
  Any Headache, Dose 2: number analyzed (Participants) | 208 | 211
  Any Headache, Dose 2 | 62 | 66
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Headache, Dose 2 | 2 | 3
  Related Headache, Dose 2: number analyzed (Participants) | 208 | 211
  Related Headache, Dose 2 | 57 | 58
  Any Myalgia, Dose 2: number analyzed (Participants) | 208 | 211
  Any Myalgia, Dose 2 | 61 | 53
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Myalgia, Dose 2 | 6 | 5
  Related Myalgia, Dose 2: number analyzed (Participants) | 208 | 211
  Related Myalgia, Dose 2 | 56 | 51
  Any Shivering, Dose 2: number analyzed (Participants) | 208 | 211
  Any Shivering, Dose 2 | 36 | 26
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Shivering, Dose 2 | 4 | 3
  Related Shivering, Dose 2: number analyzed (Participants) | 208 | 211
  Related Shivering, Dose 2 | 34 | 24
  Any Fever, Dose 2: number analyzed (Participants) | 208 | 211
  Any Fever, Dose 2 | 26 | 19
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 208 | 211
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 208 | 211
  Related Fever, Dose 2 | 24 | 18

5. Primary Outcome: Number of Days With Solicited General Symptoms
Description: Solicited general symptoms were assessed during the 7-day (Days 0-6) period after each dose.
Time Frame: During the 7-day (Days 0-6) period after each dose.
Population: The analysis was performed on subjects with solicited general symptoms from the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented and who had their symptom sheets filled in.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 91 | 93
Days
  Any Fatigue, Dose 1: number analyzed (Participants) | 69 | 59
  Any Fatigue, Dose 1 | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Any Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 31 | 14
  Any Gastrointestinal symptoms, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Any Headache, Dose 1: number analyzed (Participants) | 41 | 44
  Any Headache, Dose 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Any Myalgia, Dose 1: number analyzed (Participants) | 47 | 42
  Any Myalgia, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Any Shivering, Dose 1: number analyzed (Participants) | 25 | 17
  Any Shivering, Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Any Temperature, Dose 1: number analyzed (Participants) | 15 | 17
  Any Temperature, Dose 1 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Any Fatigue, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 30 | 27
  Any Gastrointestinal symptoms, Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Any Headache, Dose 2: number analyzed (Participants) | 62 | 66
  Any Headache, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Any Myalgia, Dose 2: number analyzed (Participants) | 61 | 53
  Any Myalgia, Dose 2 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Any Shivering, Dose 2: number analyzed (Participants) | 36 | 26
  Any Shivering, Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Any Temperature, Dose 2: number analyzed (Participants) | 26 | 19
  Any Temperature, Dose 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

6. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Symptoms (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) period after each dose.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 215 | 215
Participants
  Any AEs | 81 | 54
  Grade 3 AEs | 14 | 5
  Related AEs | 13 | 13

7. Primary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. Related SAE = SAE assessed by the investigator as related to the vaccination.
Time Frame: From first vaccination (Month 0) up to 30 days post last vaccination (Month 3)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 215 | 215
Participants
  Any SAEs | 4 | 4
  Related SAEs | 0 | 0

8. Primary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first vaccination (Month 0) up to 30 days post last vaccination (Month 3)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 215 | 215
Participants | 2 | 1

9. Secondary Outcome: Anti-gE Ab Concentrations
Description: VZV gE IgG antibody concentrations were determined by ELISA. Concentrations are presented as geometric mean concentrations (GMCs), expressed in milliinternational units per millilitre (mIU/mL).
Time Frame: At Months 0, 1, 3 and 14.
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria, who complied with the protocol requirements and for whom immunogenicity measures were available up to Month 14.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 204 | 204
mIU/mL
  At Month 0: number analyzed (Participants) | 204 | 202
  At Month 0 | 1784.3 [1572.9 to 2024.1] | 1408.5 [1203.3 to 1648.8]
  At Month 1: number analyzed (Participants) | 204 | 202
  At Month 1 | 29959.0 [26633.6 to 33699.6] | 25233.7 [22072.3 to 28848.0]
  At Month 3 | 49327.2 [45388.2 to 53608.1] | 51618.5 [47224.8 to 56420.9]
  At Month 14: number analyzed (Participants) | 197 | 199
  At Month 14 | 17783.6 [16077.1 to 19671.4] | 15784.1 [14180.2 to 17569.4]

10. Secondary Outcome: Frequencies of gE-specific Cluster of Differentiation 4 (CD4+) T-cells
Description: gE-specific CD4+ T-cells, expressing at least two activation markers (from among interferon gamma [IFN-γ], interleukin-2 [IL-2], tumour necrosis factor alpha [TNF-α] and cluster of differentiation 40-ligand [CD40L]), as determined by in vitro Intracellular Cytokine Staining (ICS).
Time Frame: At Months 0, 1, 3 and 14.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/million T-cells
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 177 | 177
CD4+ T-cells/million T-cells
  At Month 0: number analyzed (Participants) | 152 | 140
  At Month 0 | 89.09 (99.73) | 90.88 (97.5)
  At Month 1: number analyzed (Participants) | 177 | 170
  At Month 1 | 562.17 (532.58) | 534.57 (523.97)
  At Month 3: number analyzed (Participants) | 170 | 177
  At Month 3 | 2946.02 (2088.48) | 2843.89 (2111.54)
  At Month 14: number analyzed (Participants) | 103 | 148
  At Month 14 | 1290.98 (1181.89) | 1126.44 (1012.28)

11. Secondary Outcome: Number of Subjects With Any and Related SAEs
Description: as for outcome 7
Time Frame: From 30 days post last vaccination (Month 3) until study end at Month 14
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 215 | 215
Participants
  Any SAEs | 15 | 18
  Related SAEs | 0 | 0

12. Secondary Outcome: Number of Subjects With Any pIMDs
Description: as for outcome 8
Time Frame: From 30 days post last vaccination (Month 3) until study end at Month 14
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Control Group
Number analyzed (Participants) | 215 | 215
Participants | 1 | 3

ADVERSE EVENTS:
Time Frame: Solicited local and general AEs were assessed during a 7-day follow-up period (Days 0-6) after each vaccination visit. Unsolicited AEs were assessed for a period of 30 days (Days 0-29) after each vaccination visit. SAEs were assessed from the first receipt of the study vaccine (Month 0) up to study end (Month 14).
Arm/Group | GSK1437173A Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/215 | 3/215
Serious Adverse Events (participants affected / at risk) | 18/215 | 22/215
Other Adverse Events (participants affected / at risk) | 199/215 | 197/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=215) | Control Group (N=215)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (2) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=215) | Control Group (N=215)
Chills (General disorders) | 51 (61) | 37 (44)
Erythema (Skin and subcutaneous tissue disorders) | 96 (138) | 73 (101)
Fatigue (General disorders) | 114 (162) | 111 (152)
Gastrointestinal disorder (Gastrointestinal disorders) | 49 (61) | 38 (41)
Headache (Nervous system disorders) | 80 (105) | 89 (111)
Myalgia (Musculoskeletal and connective tissue disorders) | 82 (109) | 78 (96)
Pain (General disorders) | 189 (334) | 181 (321)
Pyrexia (General disorders) | 36 (41) | 32 (36)
Swelling (General disorders) | 50 (58) | 37 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.